CLINICAL TRIAL: NCT01379508
Title: OPTIMA: A Randomized, Open-label, 156-week Treatment Study to Evaluate the Efficacy and Safety of Telbivudine or Tenofovir Treatment in HBeAg-negative Chronic Hepatitis B Patients Based on the Roadmap Concept
Brief Title: Telbivudine or Tenofovir Treatment in HBeAg-negative Chronic Hepatitis B Patients Based on the Roadmap Concept
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLDT600A2409; 2007-000180-13 (Registry Identifier: Eudract)
Record Dates: First submitted 2011-06-21; First posted 2011-06-23 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-03

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Telbivudine; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- telbivudine (Experimental): telbivudine 600 mg tablet orally (p.o.) once daily for up to 156 weeks. Patients with HBV DNA ≥ 300 copies/mL at Week 24 were to initiate add-on therapy with tenofovir 300 mg tablets p.o. once daily for the remaining weeks of treatment. The investigator was to initiate tenofovir add-on therapy within 2 weeks of central laboratory confirmation. Patients with HBV DNA < 300 copies/mL at Week 24 were to continue to receive telbivudine monotherapy
  Interventions: Drug: telbivudine
- tenofovir (Active Comparator): tenofovir 300 mg tablets p.o. once daily for up to 156 weeks. Patients with HBV DNA ≥ 300 copies/mL at Week 24 were to initiate add-on therapy with telbivudine 600 mg tablet p.o. once daily for the remaining weeks of treatment. The investigator was to initiate telbivudine add-on therapy within 2 weeks of central laboratory confirmation. Patients with HBV DNA < 300 copies/mL at Week 24 were to continue to receive tenofovir monotherapy
  Interventions: Drug: tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: telbivudine — 600 mg film-coated tablets taken as 600 mg once daily
  Other Names: LDT600
  Arms: telbivudine
Drug: tenofovir disoproxil fumarate — 300 mg tablets taken as 300 mg once daily
  Arms: tenofovir

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety following the Roadmap Concept strategy with an initial monotherapy using either telbivudine or tenofovir in HBeAg negative CHB patients. The data from the study should allow for the validation of the Roadmap concept in a prospective manner, for both telbivudine and tenofovir treated HBeAg negative CHB patients. As part of a post-approval commitment to the European Health Authorities, the data will also be used to provide an optimized clinical treatment strategy for better clinical use of telbivudine in European HBeAg negative patients. Furthermore, the data from the study will contribute to a better scientific understanding, disease management and treatment of HBeAg negative CHB patients.

ELIGIBILITY:
Inclusion Criteria:

Male or female, at least 18 years of age

Documented compensated HBeAg negative CHB defined by all of the following:

* Detectable serum HBsAg at screening visit and at least 6 months prior;
* HBeAg negative at the screening visit with positive HBeAb;
* Serum HBV DNA > 2000 IU/mL Serum ALT level > 1×ULN and <10×ULN at screening visit; patient with normal ALT ≤1xULN at screening are eligible, with moderate liver inflammation or fibrosis, complensated liver sirrhosis, ALT level >1xULN wtihin last 6 months

Exclusion Criteria:

* Co-infected with HCV, HDV or HIV.
* Received treatment of nucleoside or nucleotide drugs at any time
* Received IFN or other immunomodulatory treatment within six months before Screening
* Pregnant or nursing (lactating) women
* Clinical signs/symptoms of hepatic decompensation
* History of myopathy, myositis or persistent muscle weakness
* history of clinical and laboratory evidence of chronic renal insufficency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2011-03-21 (Actual); Primary Completion 2015-12-10 (Actual); Study Completion 2015-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (25):
- Austria (2):
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Vienna
- Bulgaria (2):
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Germany (7):
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Würzburg
- Greece (4):
  - Novartis Investigative Site, Alexandroupoli, Evros
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
- Novartis Investigative Site, Caserta, CE, Italy
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Tarragona, Catalonia
  - Novartis Investigative Site, Majadahonda, Madrid
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Diyarbakır
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Trabzon

RESULTS

PARTICIPANT FLOW:
Groups:
- LdT Mono at Week 24: Patients who were initially treated with telbivudine and had hepatitis B virus deoxyribonucleic acid < 300 copies/mL in their blood at Week 24 and continued to receive 600 mg telbivudine daily after Week 24
- LdT+TDF at Week 24: Patients who were initially treated with telbivudine and had hepatitis B virus deoxyribonucleic acid > 300 copies/mL in their blood at Week 24 and continued to receive 600 mg telbivudine daily and additional 300 mg tenofovir after Week 24.
- TDF Mono at Week 24: Patients who were initially treated with tenofovir and had hepatitis B virus deoxyribonucleic acid < 300 copies/mL in their blood at Week 24 and continued to receive 300 mg tenofovir daily after Week 24.
- TDF + LdT at Week 24: Patients who were initially treated with tenofovir and had hepatitis B virus deoxyribonucleic acid > 300 copies/mL in their blood at Week 24 and continued to receive 300 mg tenofovir and additional 600 mg telbivudine after Week 24.
Period: Treatment to Week 104
Arm/Group | LdT Mono at Week 24 | LdT+TDF at Week 24 | TDF Mono at Week 24 | TDF + LdT at Week 24
Started | 99 | 22 | 109 | 11
Completed Wk 24 | 93 | 22 | 107 | 11
Treatment Exposure ≥ 52 Weeks | 91 | 21 | 105 | 11
Completed | 80 | 19 | 96 | 11
Not Completed | 19 | 3 | 13 | 0
Not completed — Adverse Event | 2 | 0 | 5 | 0
Not completed — Abnormal lab value | 1 | 0 | 0 | 0
Not completed — Abnormal test procedure result(s) | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 1 | 4 | 0
Not completed — Lost to Follow-up | 5 | 0 | 3 | 0
Not completed — Administrative problems | 3 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 1 | 0
Period: Extension Period Weeks 109-156
Arm/Group | LdT Mono at Week 24 | LdT+TDF at Week 24 | TDF Mono at Week 24 | TDF + LdT at Week 24
Started | 64 | 17 | 79 | 10
Completed | 45 | 14 | 65 | 10
Not Completed | 19 | 3 | 14 | 0
Not completed — Withdrawal by Subject | 8 | 1 | 8 | 0
Not completed — Lost to Follow-up | 6 | 1 | 5 | 0
Not completed — Administrative problems | 3 | 0 | 1 | 0
Not completed — Protocol Violation | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- LdT Mono at Week 24: Patients who had hepatitis B virus deoxyribonucleic acid < 300 copies/mL in their blood at Week 24 continued to receive 600 mg telbivudine daily after Week 24
- Total: Total of all reporting groups
Arm/Group | LdT Mono at Week 24 | LdT+TDF at Week 24 | TDF Mono at Week 24 | TDF + LdT at Week 24 | Total
Number analyzed (Participants) | 99 | 22 | 109 | 11 | 241
Age, Customized [Count of Participants; unit: Participants]
  < 30 years | 17 | 4 | 18 | 0 | 39
  Between 30 and 50 years | 56 | 13 | 59 | 7 | 135
  > 50 years | 26 | 5 | 32 | 4 | 67
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 7 | 34 | 4 | 73
  Male | 71 | 15 | 75 | 7 | 168
HBV DNA [Mean (Standard Deviation); unit: log10 copies/mL)] | 5.887 (1.2862) | 7.769 (1.2502) | 5.838 (1.2464) | 7.938 (1.0709) | 5.887 (1.2862)
HBV DNA levels < or ≥ 7 log 10 copies/mL at baseline. [Count of Participants; unit: Participants]
  < 7 log 10 copies/mL | 81 | 4 | 83 | 3 | 171
  ≥ 7 log 10 copies/mL | 18 | 18 | 26 | 8 | 70
Participants with alanine aminotransferase (ALT) - Multiples of upper limits of normal (ULN) [Count of Participants; unit: Participants] — Serum ALT normalization is an important clinically relevant efficacy endpoint. Elevated serum ALT levels are thought to reflect underlying hepatitis disease activity (i.e. active liver inflammation). Correspondingly, ALT normalization is an accepted therapeutic goal in hepatitis studies as it is thought to reflect a substantial reduction in hepatic disease activity.Measurement at baseline.
  Participants
    ≤ 1 × ULN | 46 | 3 | 52 | 4 | 105
    > 1 × - < 2 × ULN | 35 | 7 | 27 | 5 | 74
    2 × - < 5 × ULN | 13 | 11 | 26 | 1 | 51
    5 × or more ULN | 5 | 1 | 4 | 1 | 11
Participants with aspartate aminotransferase (AST) - Multiples of upper limits of normal (ULN) [Count of Participants; unit: Participants] — Measurment at baseline.
  Participants
    ≤ 1 × ULN | 70 | 10 | 69 | 2 | 151
    > 1 × - < 2 × ULN | 14 | 7 | 23 | 7 | 51
    2 × - < 5 × ULN | 12 | 4 | 16 | 1 | 33
    5 × or more ULN | 3 | 1 | 1 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving HBV DNA < 300 Copies/mL (51 IU/mL) at Week 52 (rITT Population) -
Description: The primary objective of the study is to compare the efficacy of Roadmap-Concept-based telbivudine treatment versus Roadmap-Concept-based tenofovir treatment in HBeAg-negative CHB patients. The rate of HBV DNA < 300 copies/mL (51 IU/mL) at week 52 will be used for the comparison of the efficacy. The hypothesis is that the aggregated rate of HBV DNA < 300 copies/mL (51 IU/mL) at week 52 of Telbivudine (ARM 1) is non-inferior to Tenofovir (ARM 2). For the "treating missing as failure" analysis, patients who came for their primary endpoint Week 52 visit within the ± 7-day window but not on the exact designated day of the visit were treated as "missing data."
Time Frame: week 52
Population: Roadmap intent-to-treat (rITT) population consisted of patients in the ITT population who did not discontinue before Wk 24 and did not receive add-on. The total of the mono and combination arms were analyzed.
Measure: Number; unit: percentage of participants
Groups:
- LdT Overall: Ldt Mono and LdT + TDF combined
- TDF Overall: TDF mono and TDF + LdT combined
Arm/Group | LdT Overall | TDF Overall
Number analyzed (Participants) | 113 | 117
percentage of participants
  Missing DNA data at Wk 52=failure | 91.0 | 95.0
  Imputing +/- 7 days DNA for Wk 52 | 91.9 | 95.0
  Imputing LOCF DNA for Wk 52 | 95.4 | 99.2
  Imputing within +28d DNA for Wk 52 | 92.7 | 95.0
Statistical Analysis 1: Comparison: LdT Overall vs TDF Overall; Missing DNA data at Wk 52=failure: To evaluate the primary objective, Mantel-Haenszel weighted estimates approach (stratified by HBV DNA level (< 7 log10 copies/mL or ≥ 7 log10 copies/mL) and ALT (< 3×ULN or ≥ 3×ULN) at baseline) was employed to assess the proportion of patients (response rate) who achieve HBV DNA < 300 copies/mL after 52 weeks treatment in each treatment arm, as well as the difference in proportions (telbivudine - tenofovir arm) and the 95% CI of the difference; Test type: Non-Inferiority or Equivalence — Noninferiority was derived if the lower limit of two-sided 95% CI for the difference lied above the pre-determined non-inferiority margin (-10%); Difference in percentage = -4, 95% CI 2-sided [-10.5 to 2.5]
Statistical Analysis 2: Comparison: LdT Overall vs TDF Overall; Imputing +/- 7 days DNA for Wk 52: To evaluate the primary objective, Mantel-Haenszel weighted estimates approach (stratified by HBV DNA level (< 7 log10 copies/mL or ≥ 7 log10 copies/mL) and ALT (< 3×ULN or ≥ 3×ULN) at baseline) was employed to assess the proportion of patients (response rate) who achieve HBV DNA < 300 copies/mL after 52 weeks treatment in each treatment arm, as well as the difference in proportions (telbivudine - tenofovir arm) and the 95% CI of the difference; Test type: Non-Inferiority or Equivalence — Noninferiority was derived if the lower limit of two-sided 95% CI for the difference was above the pre-determined non-inferiority margin (-10%); Difference in percentage = -3.1, 95% CI 2-sided [-9.4 to 3.1]
Statistical Analysis 3: Comparison: LdT Overall vs TDF Overall; Imputing LOCF DNA for wk 52: d/c for non response prior to Wk 52: Treating missing as failure for patients who discontinued prior to Week 52 due to unsatisfactory therapeutic effect and imputing missing with LOCF for other patients; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in percentage = -3.8, 95% CI 2-sided [-7.9 to 0.4]
Statistical Analysis 4: Comparison: LdT Overall vs TDF Overall; Imputing within +28d DNA for wk52: d/c for non response <28 days from Wk 52:Treating missing as failure for patients who discontinued prior to Week 52 due to unsatisfactory therapeutic effect and imputing missing with the earliest available assessment within the 28-day window starting from the scheduled Week 52 date for other patients (if no such assessment is available, treated as failure); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in percentage = -2.3, 95% CI 2-sided [-8.3 to 3.8]

2. Secondary Outcome: Percentage of Patients Achieving Secondary Efficacy Endpoints (rITT)
Description: To assess the antiviral efficacy, as evaluated by the percentage of patients achieving HBV DNA <300 copies/mL (51 IU/mL), ALT normalization, HBsAg loss, HBsAg conversion, virologic breakthrough (VB) at study visit, cumulative VB by study defined study period, cumulative treatment-emergent resistance
Time Frame: week 24, 52, 104
Population: Roadmap intent-to-treat (rITT) population was analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of particiipants
Arm/Group | LdT Mono at Week 24 | LdT+TDF at Week 24 | LdT Overall | TDF Mono at Week 24 | TDF + LdT at Week 24 | TDF Overall
Number analyzed (Participants) | 92 | 21 | 113 | 106 | 11 | 117
percentage of particiipants
  HBV DNA <300 Week 24 | 98.9 [94.1 to 100.0] | 0.0 [0 to 16.1] | 80.5 [72.0 to 87.4] | 99.1 [94.9 to 100.0] | 0 [0 to 28.5] | 89.7 [82.8 to 94.6]
  HBV DNA <300 Week 104 | 69.6 [59.1 to 78.7] | 76.2 [52.8 to 91.8] | 70.8 [61.5 to 79.0] | 74.5 [65.1 to 82.5] | 81.8 [48.2 to 97.7] | 75.2 [66.4 to 82.7]
  HBV DNA <300 Week 24 LOCF | 100.0 [96.1 to 100.0] | 0 [0 to 16.1] | 81.4 [73.0 to 88.1] | 100.0 [96.6 to 100.0] | 0 [0 to 28.5] | 90.6 [83.8 to 95.2]
  HBV DNA <300 Wk104 LOCF | 92.4 [84.9 to 96.9] | 100.0 [83.9 to 100.0] | 93.8 [87.7 to 97.5] | 99.1 [94.9 to 100.0] | 100.0 [71.5 to 100.0] | 99.1 [95.3 to 100.0]
  ALT Normalization Wk 52 | 84.0 [70.9 to 92.8] | 83.3 [58.6 to 96.4] | 83.8 [72.9 to 91.6] | 82.5 [70.1 to 91.3] | 85.7 [42.1 to 99.6] | 82.8 [71.3 to 91.1]
  ALT Normalization Week 104 | 70.0 [55.4 to 82.1] | 72.2 [46.5 to 90.3] | 70.6 [58.3 to 81.0] | 61.4 [47.6 to 74.0] | 85.7 [42.1 to 99.6] | 64.1 [51.1 to 75.7]
  ALT Normalization Wk 52 LOCF | 88.0 [75.7 to 95.5] | 83.3 [58.6 to 96.4] | 86.8 [76.4 to 93.8] | 87.7 [76.3 to 94.9] | 85.7 [42.1 to 99.6] | 87.5 [76.8 to 94.4]
  ALT Normalization Wk 104 LOCF | 92.0 [80.8 to 97.8] | 83.3 [58.6 to 96.4] | 89.7 [79.9 to 95.8] | 86.0 [74.2 to 93.7] | 85.7 [42.1 to 99.6] | 85.9 [75.0 to 93.4]
  HBsAg loss Week 52 | 0 [0 to 3.9] | 0 [0 to 16.1] | 0 [0 to 3.2] | 0 [0 to 3.4] | 0 [0 to 28.5] | 0 [0 to 3.1]
  HBsAg loss Week 104 | 0 [0 to 3.9] | 0 [0 to 16.1] | 0 [0 to 3.2] | 0 [0 to 3.4] | 0 [0 to 28.5] | 0 [0 to 3.1]
  HBsAg conversion Week 52 | 0 [0 to 3.9] | 0 [0 to 16.1] | 0 [0 to 3.2] | 0 [00 to 3.4] | 0 [0 to 28.5] | 0 [0 to 3.1]
  HBsAg conversion Week 104 | 0 [0 to 3.9] | 0 [0 to 16.1] | 0 [0 to 3.2] | 0 [0 to 3.4] | 0 [0 to 28.5] | 0 [0 to 3.1]
  Cum virol break BaseL to Wk 24 | 0 [0 to 3.9] | 4.8 [0.1 to 23.8] | 0.9 [0.0 to 4.8] | 0 [0 to 3.4] | 0 [0 to 28.5] | 0 [0 to 3.1]
  Cum virol break Wk 24 to Wk 52 | 3.3 [0.7 to 9.2] | 0 [0 to 16.1] | 2.7 [0.6 to 7.6] | 0 [0 to 3.4] | 0 [0 to 28.5] | 0 [0 to 3.1]
  Cum virol break Wk 52 to Wk 104 | 12.0 [6.1 to 20.4] | 0 [0 to 16.1] | 9.7 [5.0 to 16.8] | 1.9 [0.2 to 6.6] | 0 [0 to 28.5] | 1.7 [0.2 to 6.0]
  Cum virol break BaseLto Wk 104 | 14.1 [7.7 to 23.0] | 4.8 [0.1 to 23.8] | 12.4 [6.9 to 19.9] | 1.9 [0.2 to 6.6] | 0 [0 to 28.5] | 1.7 [0.2 to 6.0]
  Cum vir break BL to Wk24 LOCF | 0 [0 to 3.9] | 4.8 [0.1 to 23.8] | 0.9 [0.0 to 4.8] | 0 [0 to 3.4] | 0 [0 to 28.5] | 0 [0 to 3.1]
  Cum virol break Wk 24 to Wk 52 LOCF | 3.3 [0.7 to 9.2] | 0 [0 to 16.1] | 2.7 [0.6 to 7.6] | 0 [0 to 3.4] | 0 [0 to 28.5] | 0 [0 to 3.1]
  Cum virol break Wk52-Wk104 LOCF | 12.0 [6.1 to 20.4] | 0 [0 to 16.1] | 9.7 [5.0 to 16.8] | 1.9 [0.2 to 6.6] | 0 [0 to 28.5] | 1.7 [0.2 to 6.0]
  Cum virol break BLto Wk 104 LOCF | 14.1 [7.7 to 23.0] | 4.8 [0.1 to 23.8] | 12.4 [6.6 to 19.9] | 1.9 [0.2 to 6.6] | 0 [0 to 28.5] | 1.7 [0.2 to 6.0]
  Cum tx emergent resistance Wk 52 | 3.3 [0.7 to 9.2] | 0 [0 to 16.1] | 2.7 [0.6 to 7.6] | 0 [0 to 3.4] | 0 [0 to 28.5] | 0 [0 to 3.1]
  Ccum tx emergent resistance Wk 104 | 9.2 [4.1 to 17.3] | 0 [0 to 16.1] | 7.4 [3.3 to 14.1] | 0 [0 to 3.5] | 0 [0 to 28.5] | 0 [0 to 3.1]
  Cum tx emergent resist Wk52 LOCF | 3.3 [0.7 to 9.2] | 0 [0 to 16.1] | 2.7 [0.6 to 7.6] | 0 [0 to 3.4] | 0 [0 to 28.5] | 0 [0 to 3.1]
  Cum tx emergent resist Wk 104 LOCF | 9.2 [4.1 to 17.3] | 0 [0 to 16.1] | 7.4 [3.3 to 14.1] | 0 [0 to 3.5] | 0 [0 to 28.5] | 0 [0 to 3.1]
  <7 log at BL HBV DNA <300 Wk52 | 93.4 [85.3 to 97.8] | 75.0 [19.4 to 99.4] | 92.5 [84.4 to 97.2] | 95.0 [87.7 to 98.6] | 100.0 [29.2 to 100.0] | 95.2 [88.1 to 98.7]
  <7 log HBV DNA <300 Wk104 | 68.4 [56.7 to 78.6] | 50.0 [6.8 to 93.2] | 67.5 [56.1 to 77.6] | 76.3 [65.4 to 85.1] | 66.7 [9.4 to 99.2] | 75.9 [65.3 to 84.6]
  <7 log HBV DNA <300 Wk 52 LOCF | 97.4 [90.8 to 99.7] | 100.0 [39.8 to 100.0] | 97.5 [91.3 to 99.7] | 100.0 [95.5 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [95.7 to 100.0]
  <7 log HBV DNA <300 Wk 104 LOCF | 92.1 [83.6 to 97.0] | 100.0 [39.8 to 100.0] | 92.5 [84.4 to 97.2] | 98.8 [93.2 to 100.0] | 100.0 [29.2 to 100.0] | 98.8 [93.5 to 100.0]

3. Secondary Outcome: Percentage of Participants Achieving Secondary Efficacy Endpoints at Week 156 (mITT)
Description: To assess the antiviral efficacy, as evaluated by the percentage of patients achieving HBV DNA <300 copies/mL (51 IU/mL) at Week156, ALT normalization, HBsAg loss, development of HBsAg conversion , cumulative tx emergent resistance, HBV DNA <300 copies/mL with HBV DNA <7 log at Baseline
Time Frame: 156 weeks
Population: The modified ITT (mITT) population consisted of all patients in ITT population who were eligible and enrolled into the extension.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LdT Mono at Week 24 | LdT+TDF at Week 24 | LdT Overall | TDF Mono at Week 24 | TDF + LdT at Week 24 | TDF Overall
Number analyzed (Participants) | 62 | 17 | 79 | 79 | 10 | 89
percentage of participants
  HBV DNA < 300 Week 156 | 17.7 [9.2 to 29.5] | 11.8 [1.5 to 36.4] | 16.5 [9.1 to 26.5] | 13.9 [7.2 to 23.5] | 20.0 [2.5 to 55.6] | 14.6 [8.0 to 23.7]
  HBV DNA < 300 Wk156 LOCF | 88.7 [78.1 to 95.3] | 100.0 [80.5 to 100.0] | 91.1 [82.6 to 96.4] | 100.0 [95.4 to 100.0] | 100.0 [69.2 to 100.0] | 100.00 [95.9 to 100.00]
  ALT normalization Wk 156 | 14.3 [4.8 to 30.3] | 6.7 [0.2 to 31.9] | 12.0 [4.5 to 24.3] | 10.5 [2.9 to 24.8] | 28.6 [3.7 to 71.0] | 13.3 [5.1 to 26.8]
  ALT normalization Wk 156 LOCF | 85.7 [69.7 to 95.2] | 93.3 [68.1 to 99.8] | 88.0 [75.7 to 95.5] | 86.8 [71.9 to 95.6] | 85.7 [42.1 to 99.6] | 86.7 [73.2 to 94.9]
  HBSAg loss/ seroconversion | 0 [0 to 5.8] | 0 [0 to 19.5] | 0 [0 to 4.6] | 0 [0 to 4.6] | 0 [0 to 30.8] | 0 [0 to 4.1]
  Cum VB Wk104-156 LOCF | 16.1 [8.0 to 27.7] | 0 [0 to 19.5] | 12.7 [6.2 to 22.0] | 1.3 [0 to 6.9] | 0 [0 to 30.8] | 1.1 [0.0 to 6.1]
  Cum VB BL to Wk 156 LOCF | 21.0 [11.7 to 33.2] | 0 [0 to 19.5] | 16.5 [9.1 to 26.5] | 1.3 [0 to 6.9] | 0 [0 to 30.8] | 1.1 [0.0 to 6.1]
  Cum tx emerg resist Week 156 LOCF | 14.0 [6.3 to 25.8] | 0 [0 to 19.5] | 10.8 [4.8 to 20.2] | 0 [0 to 4.6] | 0 [0 to 30.8] | 0 [0 to 4.1]
  HBV DNA < 300 Wk156 <7 log at BL | 17.6 [8.4 to 30.9] | 0 [0 to 70.8] | 16.7 [7.9 to 29.3] | 11.7 [4.8 to 22.6] | 50.0 [1.3 to 98.7] | 12.9 [5.7 to 23.9]
  HBV DNA <300 Wk156 <7 log LOCF | 88.2 [76.1 to 95.6] | 100.0 [29.2 to 100.0] | 88.9 [77.4 to 95.8] | 100.0 [94.0 to 100.0] | 100.0 [15.8 to 100.0] | 100.0 [94.2 to 100.0]
  Cum tx-emerg resist Wk156 <7log LOCF | 8.7 [2.4 to 20.8] | 0.0 [0.0 to 70.8] | 8.2 [2.3 to 19.6] | 0.0 [0.0 to 6.0] | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 5.8]

4. Secondary Outcome: eGFR Change From Baseline in Telbivudine Arm vs Tenofovir Arm Over the Course of the Study
Description: eGFR changes were calculated using the Modification of Diet in Renal Disease (MDRD) formula: GFR = 186 x (sCr)^(-1.154) x (age)^-0.203 with Female: Multiply GFR by 0.742; Black: Multiply GFR by 1.210. sCr is Serum Creatinine in mg/dl (measured at each scheduled visit). Age in years at visit (=[sCr sample collection date -Date of birth]/365.25). Weight in kilograms, as measured at the visit or the closest previous visit Safety population.
Time Frame: Baseline, 24 weeks, 52 weeks, 104 weeks, 156 weeks
Population: Safety population consisted of patients who received at least 1 dose of study drug and had 1 post-baseline safety assessment. Numbers in parentheses represent the number of participants who met the criteria for the measurement in the 2 LDT arms, LDT Overall, 2 TDF arms, TDF Overall, respectively
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m2
Arm/Group | LdT Mono at Week 24 | LdT+TDF at Week 24 | LdT Overall | TDF Mono at Week 24 | TDF + LdT at Week 24 | TDF Overall
Number analyzed (Participants) | 98 | 22 | 120 | 109 | 11 | 120
mL/min/1.73 m2
  Week 24 change (97,22,119,108,11,119) | 1.43 (12.815) | -12.06 (14.394) | -1.07 (14.076) | -2.41 (14.885) | -7.17 (15.368) | -2.85 (14.928)
  Week 52 change(97,22,119,108,11,119) | 5.18 (18.842) | -6.80 (17.229) | 2.96 (19.064) | -2.70 (18.636) | -8.39 (10.479) | -3.22 (18.082)
  Week 104 change(97,22,119,108,11,119) | 5.19 (16.583) | -5.77 (15.943) | 3.16 (16.947) | -3.83 (15.157) | -8.69 (15.632) | -4.28 (15.200)
  Week 156 change(62,17,79,79,10,89) | 8.07 (16.777) | -10.89 (14.993) | 3.99 (18.104) | -5.34 (13.393) | -6.67 (11.905) | -5.49 (13.178)
  Baseline actual(98,22,120,109,11,120) | 94.71 (16.422) | 109.79 (19.560) | 97.47 (17.936) | 95.91 (16.396) | 94.50 (17.558) | 95.78 (16.433)
  Week 24 actual(97,22,119,108,11,119) | 96.43 (16.434) | 97.73 (17.690) | 96.67 (16.603) | 93.61 (18.500) | 87.33 (16.854) | 93.03 (18.378)
  Week 52 actual(97,22,119,108,11,119) | 100.18 (20.257) | 102.99 (19.425) | 100.70 (20.054) | 93.32 (18.880) | 86.12 (14.233) | 92.66 (18.569)
  Week 104 actual (97,22,119,108,11,119) | 100.20 (16.287) | 104.02 (18.201) | 100.90 (16.643) | 92.19 (18.240) | 85.81 (13.099) | 91.60 (17.879)
  Week 156 actual(62,17,79,79,10,89) | 101.33 (18.505) | 100.70 (20.029) | 101.20 (18.712) | 88.83 (16.773) | 87.93 (13.280) | 88.73 (16.355)

ADVERSE EVENTS:
Groups:
- LdT Mono at Week 24: LdT Mono at Week 24
- LdT + TDF at Week 24: LdT + TDF at Week 24
- TDF Mono at Week 24: TDF Mono at Week 24
- TDF + LdT at Week 24: TDF + LdT at Week 24
Arm/Group | LdT Mono at Week 24 | LdT + TDF at Week 24 | TDF Mono at Week 24 | TDF + LdT at Week 24
Serious Adverse Events (participants affected / at risk) | 6/98 | 5/22 | 11/109 | 2/11
Other Adverse Events (participants affected / at risk) | 60/98 | 15/22 | 56/109 | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LdT Mono at Week 24 (N=98) | LdT + TDF at Week 24 (N=22) | TDF Mono at Week 24 (N=109) | TDF + LdT at Week 24 (N=11)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Gastroduodenitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 3 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 3 | 0
Metastases to abdominal wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Psychogenic pain disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LdT Mono at Week 24 (N=98) | LdT + TDF at Week 24 (N=22) | TDF Mono at Week 24 (N=109) | TDF + LdT at Week 24 (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 6 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 6 | 0 | 5 | 3
Diarrhoea (Gastrointestinal disorders) | 8 | 0 | 5 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 0 | 5 | 1
Gastritis (Gastrointestinal disorders) | 6 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 10 | 3 | 2 | 3
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Asthenia (General disorders) | 5 | 1 | 0 | 2
Fatigue (General disorders) | 5 | 1 | 8 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 1 | 2
Pyrexia (General disorders) | 1 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 1
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 8 | 2 | 8 | 2
Nasopharyngitis (Infections and infestations) | 7 | 2 | 8 | 1
Respiratory tract infection (Infections and infestations) | 3 | 0 | 1 | 1
Rhinitis (Infections and infestations) | 5 | 2 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 5 | 0 | 5 | 1
Amylase increased (Investigations) | 1 | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 7 | 1 | 4 | 0
Blood creatine phosphokinase increased (Investigations) | 24 | 10 | 17 | 2
Blood phosphorus increased (Investigations) | 1 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 8 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 2 | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 2
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 17 | 3 | 16 | 2
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1
Crystalluria (Renal and urinary disorders) | 0 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 5 | 1 | 0
Nephroptosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 7 | 4 | 5 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No